CLINICAL TRIAL: NCT03765502
Title: A Simulation Study Comparing Successful Administration, Time to Administer, and User Experience of Ready-to-Use Nasal Glucagon With Reconstitutable Injectable Glucagon
Brief Title: A Study Comparing User Experience of Different Delivery Devices for Glucagon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17156; I8R-MC-IGBM (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-11-16; First posted 2018-12-05 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2019-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Nasal Glucagon Device (NG) (Experimental): Empty NG device administered to a manikin during simulations of severe hypoglycaemia emergencies. No drug will be administered to humans.
  Interventions: Device: Nasal Glucagon Device (NG)
- Glucagon Emergency Kit (GEK) (Active Comparator): Commercially available GEK delivered intramuscularly to a manikin during simulations of severe hypoglycaemia emergencies. No drug will be administered to humans.
  Interventions: Device: GEK; Drug: IM Glucagon

INTERVENTIONS:
Device: Nasal Glucagon Device (NG) — NG devices will be provided empty of drug product
  Arms: Nasal Glucagon Device (NG)
Device: GEK — Used to administer glucagon intramuscularly (IM)
  Arms: Glucagon Emergency Kit (GEK)
Drug: IM Glucagon — Administered IM via GEK
  Arms: Glucagon Emergency Kit (GEK)

SUMMARY:
The purpose of the study is to learn more about different devices for delivering glucagon during simulations of severe hypoglycemic (low blood sugar) emergencies. The study will be carried out using medical manikins to simulate real life scenarios. No drug will be administered to humans. Part A will last approximately 17 days for Trained Users and Participants with Diabetes (PWD). Part B will last approximately nine (9) days for Untrained Users. Each part will be separated by approximately 7 days.

ELIGIBILITY:
Inclusion Criteria:

All participants (Trained Users, Participants with Diabetes [PWDs] and Untrained Users):

* Are able to understand the purpose and procedure of the study and to give written informed consent to show willingness to participate in the study

Trained Users only:

* Are participants who are not diagnosed with Type 1 Diabetes Mellitus (T1DM) or Type 2 Diabetes Mellitus (T2DM)
* Are close friends/relatives of a patient with T1DM or T2DM on insulin
* Have not previously administered any rescue medications (e.g. epinephrine, glucagon, narcan or seizure medications)

Untrained Users only:

* Have not been diagnosed with T1DM or T2DM, and are not a Trained User of a person with T1DM or T2DM
* Have not previously administered any rescue medications (e.g. epinephrine, glucagon, narcan or seizure medications)

Exclusion Criteria:

All participants (Trained Users, PWDs and Untrained Users):

* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Trained Users and Untrained Users only (i.e. the participants involved in the simulations):

* Are currently enrolled in a clinical study involving any type of medical research judged not to be scientifically or medically compatible with this study
* Are judged by the investigator as being likely to have difficulty performing the administration due to physical, cognitive and/or severe psychiatric disorder
* Are judged by the investigator as being trained or experienced in performing rescue drug administration
* Are judged by the investigator as being trained or experienced in performing high-fidelity simulations of drug administration
* Have received formal training in a medical field, and/or worked in this field within the prior 5 years; or otherwise are judged by the investigator as being trained or experienced as a first responder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trained Users were recruited alongside a participant with diabetes (PWD) with whom they were familiar. They were given a level of training intended to mimic that of a real-life caregiver on both devices: glucagon emergency kit (GEK) and nasal glucagon (NG). Untrained Users who have limited knowledge of severe hypoglycemia did not receive training.
Pre-assignment Details: Trained users participated in Part A and untrained users participated in Part B.
Groups:
- Part A Trained Users NG/GEK: Simulation 1: Day 8 participants were trained to administer an empty nasal glucagon device to a manikin during a simulation of severe hypoglycemia emergency.
  Simulation 2: Day 15 participants were trained to administer a glucose emergency kit intramuscularly to a manikin during a simulation of severe hypoglycemia emergency.
  No drug was administered to humans in either simulation.
- Part A Trained Users GEK/NG: Simulation 1: Day 8 participants were trained to administer a glucose emergency kit intramuscularly to a manikin during a simulation of severe hypoglycemia emergency.
  Simulation 2: Day 15 participants were trained to administer an empty nasal glucagon device to a manikin during a simulation of severe hypoglycemia emergency.
  No drug was administered to humans in either simulation.
- Part A Person With Diabetes (PWD): Day 1 - PWD trained participants to administer a glucose emergency kit intramuscularly or an empty nasal glucagon device (depending on randomization).
  Simulation 1: Day 8 - PWD trained participants to administer an empty nasal glucagon device or a glucose emergency kit intramuscularly(depending on randomization).
  No drug was administered to humans in either simulation.
- Part B Untrained Users NG/GEK: Simulation1: Day 1 untrained participants administered an empty nasal glucagon device to a manikin during a simulation of severe hypoglycemia emergency.
  Simulations 2: Day 8 untrained participants administered a glucose emergency kit intramuscularly to a manikin during a simulation of severe hypoglycemia emergency.
  No drug was administered to humans in either simulation.
- Part B Untrained Users GEK/NG: Simulation 1: Day 1 untrained participants administered a glucose emergency kit intramuscularly to a manikin during a simulation of severe hypoglycemia emergency.
  Simulation 2: Day 8 untrained participants administered an empty nasal glucagon device to a manikin during a simulation of severe hypoglycemia emergency.
  No drug was administered to humans in either simulation.
Period: Simulation 1
Arm/Group | Part A Trained Users NG/GEK | Part A Trained Users GEK/NG | Part A Person With Diabetes (PWD) | Part B Untrained Users NG/GEK | Part B Untrained Users GEK/NG
Started | 20 | 13 | 33 | 16 | 17
Completed | 20 | 13 | 33 | 16 | 17
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Simulation 2
Arm/Group | Part A Trained Users NG/GEK | Part A Trained Users GEK/NG | Part A Person With Diabetes (PWD) | Part B Untrained Users NG/GEK | Part B Untrained Users GEK/NG
Started | 20 | 12 (Participant completed Period 1 GEK simulation but did not return for the Period 2 NG simulation.) | 32 (PWD completed Period 1 GEK simulation but did not return for the Period 2 NG simulation.) | 16 | 17
Completed | 20 | 12 | 32 | 16 | 17
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized trained user participants, untrained user participants, and participants with diabetes.
Groups:
- Part A Trained Users: All trained participants in Part A
- Part A Participants With Diabetes: All participants with diabetes in Part A
- Part B Untrained Users: All participants in Part B.
- Total: Total of all reporting groups
Arm/Group | Part A Trained Users | Part A Participants With Diabetes | Part B Untrained Users | Total
Number analyzed (Participants) | 33 | 33 | 33 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 32 | 33 | 94
  >=65 years | 4 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 15 | 60
  Male | 10 | 11 | 18 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 17 | 13 | 47
  White | 13 | 15 | 18 | 46
  More than one race | 2 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 33 | 33 | 99

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Trained Users That Performed a Successful Administration for Each Device
Description: Percentage of trained users who found both devices and performed a successful administration of both rescue devices for both simulations.
Time Frame: Part A: Days 8 - 9 and Days 15 - 17
Population: All trained user participants who found both devices and participated in at least one simulation of a rescue device. Participants with diabetes (PWD) reporting group data not collected per protocol.
Measure: Number; unit: percentage of participants
Groups:
- Nasal Glucagon (NG): Trained participants who found and had a successful administration of NG rescue device.
- Glucagon Emergency Kit (GEK): Trained participants who found had a successful administration of the GEK rescue device.
Arm/Group | Nasal Glucagon (NG) | Glucagon Emergency Kit (GEK)
Number analyzed (Participants) | 31 | 32
percentage of participants | 90.3 | 15.6
Statistical Analysis 1: Comparison: Nasal Glucagon (NG) vs Glucagon Emergency Kit (GEK); Test type: Superiority; p < .0001, McNemar; Crossover design: paired test

2. Secondary Outcome: Percentage of Untrained Users That Perform a Successful Administration for Each Device
Description: Percentage of untrained users who found both devices and performed a successful administration of both rescue devices for both simulations.
Time Frame: Part B: Day 1 and Days 8-9
Population: All untrained user participants who found both devices and participated in at least one simulation of a rescue device.
Measure: Number; unit: percentage of participants
Groups:
- Nasal Glucagon (NG): Participants who were not trained on the administration of NG rescue device.
- Glucagon Emergency Kit (GEK): Participants who were not trained on the administration of the GEK.
Arm/Group | Nasal Glucagon (NG) | Glucagon Emergency Kit (GEK)
Number analyzed (Participants) | 33 | 31
percentage of participants | 90.9 | 0
Statistical Analysis 1: Comparison: Nasal Glucagon (NG) vs Glucagon Emergency Kit (GEK); Test type: Superiority; p < .0001, McNemar; Crossover design: paired test

3. Secondary Outcome: Average Time for Trained Users to Successfully Administer One Device Over the Other
Description: Average time for trained users who found both devices to successfully administer one rescue device over the other in Part A.
Time Frame: Part A: Day 8 and Days 15-17
Population: All trained user participants who found both devices and completed at least one device simulation. PWD reporting group data not collected per protocol.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Nasal Glucagon (NG): Trained participants who found device and had a successful administration of NG rescue device.
- Glucagon Emergency Kit (GEK): Trained participants who found device and had a successful administration of GEK rescue device.
Arm/Group | Nasal Glucagon (NG) | Glucagon Emergency Kit (GEK)
Number analyzed (Participants) | 28 | 32
seconds | 47.3 (52.0) | 81.8 (18.6)

4. Secondary Outcome: Average Time for Untrained Users to Successfully Administer One Device Over the Other
Description: Average time for untrained users who found both devices to successfully administer one rescue device over the other in Part B. To successfully administer either NG or GEK, a participant must complete all of the critical steps for each device, and administer a complete dose.
Time Frame: Part B: Day 1 and Days 8-9
Population: All untrained user participants who found both devices and completed at least one successful rescue device simulation.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Nasal Glucagon Device (NG): Untrained participants who found device and had a successful administration of NG rescue device.
- Glucagon Emergency Kit (GEK): Untrained participants who found device and had a successful administration of GEK rescue device.
Arm/Group | Nasal Glucagon Device (NG) | Glucagon Emergency Kit (GEK)
Number analyzed (Participants) | 30 | 33
seconds | 44.5 (47.8) | NA (NA) — There were no successful administrations of the Glucagon Emergency Kit for the untrained participants. Data for average time of unsuccessful administrations were not collected.

5. Secondary Outcome: Percentage of Participants (Trained and Untrained Users) That Prefer One Device Over the Other
Description: Overall preference was measured via the Rescue Device Preference (RDP) questionnaire completed by Trained and Untrained participant users. Participants rated their preference for NG or GEK by choosing one of five radio buttons: Strongly prefer NG, prefer NG, no preference, prefer GEK, strongly prefer GEK. Data here represents pooling for Part A and Part B.
Time Frame: Part A: Days 8-9; Day 15-17 and Part B: Day 1; Days 8-9
Population: All trained and untrained participants who found both devices and completed the rescue device preference questionnaire for Part A and Part B combined. PWD reporting group data not collected per protocol.
Measure: Number; unit: percentage of participants
Groups:
- Part A (Trained): Overall preference for Trained users (Part A) for rescue device, NG and GEK.
- Part B (Untrained): Overall preference for Untrained users (Part B) for rescue device, NG and GEK.
Arm/Group | Part A (Trained) | Part B (Untrained)
Number analyzed (Participants) | 31 | 31
percentage of participants
  Strongly Prefer Nasal Glucagon | 58.1 | 71.0
  Prefer Nasal Glucagon | 22.6 | 22.6
  No Preference | 6.5 | 3.2
  Prefer Injectable Glucagon | 6.5 | 0.0
  Strongly Prefer Injectable Glucagon | 6.5 | 3.2

6. Secondary Outcome: Percentage of Participants (PWD) That Prefer One Device Over the Other
Description: Preference was measured by the PWD overall feeling of being safer during a severe low blood sugar event using Rescue Device Preference-Associated Person (RDP-AP). Participants rated their preference for NG or GEK by choosing one of five radio buttons: Strongly prefer NG, prefer NG, no preference, prefer GEK, strongly prefer GEK.
Time Frame: Part A: Days 15 - 17
Population: All PWD who completed the device preference questionnaire.
Measure: Number; unit: percentage of participants
Groups:
- Participant With Diabetes (PWD): Preference was measured by the PWD overall feeling of being safer during a severe low blood sugar event using Rescue Device Preference-Associated Person (RDP-AP). Participants rated their preference for NG or GEK by choosing one of five radio buttons: Strongly prefer NG, prefer NG, no preference, prefer GEK, strongly prefer GEK.
Arm/Group | Participant With Diabetes (PWD)
Number analyzed (Participants) | 32
percentage of participants
  Strongly Prefer Nasal Glucagon | 78.1
  Prefer Nasal Glucagon | 12.5
  No Preference | 3.1
  Prefer Injectable Glucagon | 0.0
  Strongly Prefer Injectable Glucagon | 6.3

7. Secondary Outcome: Percentage of Participants Trained and Untrained Users That Find One Device Easy to Use Over the Other
Description: Ease of use was measured via the Individual Rescue Device Ease of Use (RDEU) Questionnaire by Trained and Untrained Participants. Participants answered three questions about ease of use for each device by choosing one of five radio buttons: Strongly disagree, disagree, neither disagree nor agree, agree, strongly agree. Data here represents pooling of Simulation 1 for Part A and Part B.
Time Frame: Part A: Days 15 -17 and Part B: Days 8 - 9
Population: All trained and untrained users who found both devices and completed the device preference questionnaires. PWD reporting group data not collected per protocol.
Measure: Number; unit: percentage of participants
Groups:
- Part A (Trained): Overall ease of use for Trained users (Part A) for rescue device, NG and GEK.
- Part B (Untrained): Overall ease of use for Untrained users (Part B) for rescue device, NG and GEK.
Arm/Group | Part A (Trained) | Part B (Untrained)
Number analyzed (Participants) | 31 | 31
percentage of participants
  Strongly Prefer Nasal Glucagon | 48.4 | 80.6
  Prefer Nasal Glucagon | 29.0 | 16.1
  No Preference | 9.7 | 0.0
  Prefer Injectable Glucagon | 6.5 | 0.0
  Strongly Prefer Injectable Glucagon | 3.2 | 3.2

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 17 days)
Description: All participants who participated in at least one training or simulation of a study device.
Groups:
- Part A Trained Users Nasal Glucagon (NG): Trained users NG.
- Part A Trained Users Glucagon Emergency Kit (GEK): Trained user GEK.
- Part A Participants With Diabetes (PWD): PWD
- Part B Untrained Users NG: Untrained user NG.
- Part B Untrained Users GEK: Untrained user GEK.
Arm/Group | Part A Trained Users Nasal Glucagon (NG) | Part A Trained Users Glucagon Emergency Kit (GEK) | Part A Participants With Diabetes (PWD) | Part B Untrained Users NG | Part B Untrained Users GEK
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32 | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32 | 0/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32 | 0/33 | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The agreement also provides that if CRU is unwilling to delay the publication or presentation, CRU will remove the information which sponsor has specified it reasonably believes would jeopardize its intellectual property interests.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT03765502/SAP_000.pdf
  • Study Protocol (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT03765502/Prot_001.pdf